CLINICAL TRIAL: NCT02458092
Title: Phase 1b Controlled Double Blind Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of the Candidate Plasmodium Falciparum Malaria Protein 010 (FMP010) Administered Intramuscularly With Glaxo Smith Kline (GSK) Biologicals' Adjuvant AS01B
Brief Title: Evaluate the Safety and Efficacy of Plasmodium Falciparum Malaria Protein 010 (FMP010) Administered With Adjuvant AS01B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); United States Agency for International Development (USAID) (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A-14620.b; WRAIR 1417 (Other: Walter Reed Army Institute of Research)
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 50 µg of FMP010 antigen in 0.5 mL AS01B adjuvant (Experimental): 50 µg of FMP010 antigen in 0.5 mL AS01B adjuvant given intramuscularly in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Plasmodium falciparum Malaria Protein 010 (FMP010)
- Rabies Vaccine Rabipur (Experimental): Rabies Vaccine Rabipur given intramuscularly in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Rabipur

INTERVENTIONS:
Biological: Plasmodium falciparum Malaria Protein 010 (FMP010) — Vaccine antigen is a recombinant protein based on merozoite surface protein-1 (MSP-1) of FVO strain of Plasmodium falciparum, and adjuvant AS01B is a proprietary adjuvant of GSK
  Arms: 50 µg of FMP010 antigen in 0.5 mL AS01B adjuvant
Biological: Rabipur — Rabipur is a licensed rabies vaccine.
  Arms: Rabies Vaccine Rabipur

SUMMARY:
The purpose of this study is to determine whether an investigational malaria vaccine is safe and induces an immune response against malaria when tested in adults living in the United States.

DETAILED DESCRIPTION:
Study is to evaluate the safety, reactogenicity, and immunogenicity fo the candidate Plasmodium falciparum malaria protein 10 (FMP010). Malaria-experienced adults will be enrolled and randomized into 2 groups. Subjects will receive full dose FMP010 antigen (approximately 50 μg) in 0.5 mL AS01B adjuvant or licensed rabies vaccine Rabipur (by Novartis) supplied in single dose vials containing lyophilized antigen with 1.0 mL of diluent (sterile water) for injection.

ELIGIBILITY:
Inclusion Criteria:

* • A male or non-lactating female 18 to 50 years of age (inclusive) at the time of screening

  * Free of significant health problems as established by medical history and clinical examination before entering into the study
  * Available to participate for duration of study (approximately seven months)

If the subject is female, she must be of non-childbearing potential (either surgically sterilized or one year post-menopausal) or, if of childbearing potential, she must have a negative pregnancy test at the time of vaccination, be capable of preventing pregnancy for at least one month prior to determination of eligibility (to include abstinence or contraceptives (for example intrauterine contraceptive device; oral contraceptives; Norplant® or Depo-Provera® ), and must agree to continue such precautions for two months after completion of the vaccination series.

Written informed consent must be obtained from the subject before screening procedures.

Exclusion Criteria:

* • Prior receipt of any investigational malaria vaccine

  * Prior receipt of a vaccine containing either QS-21, MPL or AS02A or AS01B
  * Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period
  * Administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within six months of vaccination. For corticosteroids, this is defined as prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed.
  * Planned administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of the study vaccine.
  * Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
  * A family history of congenital or hereditary immunodeficiency
  * Chronic or active neurologic disease including seizure disorder
  * History of splenectomy
  * Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or abnormal baseline laboratory screening tests

    * ALT above normal range
    * Creatinine above normal range
    * Hemoglobin below normal range
    * Platelet count below normal range
    * Total white cell count below normal
  * Acute disease at the time of enrollment (acute disease is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness, such as diarrhea or mild upper respiratory infection without fever, i.e. Oral temperature < 37.5°C.
  * Hepatomegaly, right upper quadrant abdominal pain or tenderness
  * Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
  * Pregnant or lactating female
  * Suspected or known current alcohol abuse/drug abuse as obtained by history and physical examination
  * Female who is willing or intends to become pregnant during the study
  * Any history of allergic reaction or anaphylaxis to previous vaccination
  * Unwilling to allow blood samples to be stored for future use
  * Inability to make follow up visits
  * Allergy to kanamycin, nickel, or imidazole
  * Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study
  * Previous allergy to Rabies Vaccine
  * Allergy to chicken and chicken products

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nekoye Otsyula, Principal Investigator — US Army Medical Research Unit - Kenya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 healthy, malaria-experienced adults were enrolled and randomized into 2 groups at Walter Reed Project/Kenya Medical Research Institute (KEMRI) Kisumu, Kenya.
Groups:
- 50 ug of FMP010 Antigen in 0.5 mL AS01B Adjuvant: Plasmodium falciparum Malaria Protein 010 (FMP010): Vaccine antigen is a recombinant protein based on merozoite surface protein-1 (MSP-1) of FVO strain of Plasmodium falciparum, and adjuvant AS01B is a proprietary adjuvant of GSK. Vaccinations were performed intramuscularly in the deltoid muscle of the non-dominant arm, 3 doses were given at 0-, 1-, 2-month interval.
- Rabies Vaccine Rabipur: Rabipur: Rabipur is a licensed rabies vaccine (by Novartis) supplied in single dose vials containing lyophilized antigen with 1.0 mL of diluent (sterile water) for injection. Vaccinations were performed intramuscularly in the deltoid muscle of the non-dominant arm, 3 doses were given at 0-, 1-, 2-month interval.
Period: Overall Study
Arm/Group | 50 ug of FMP010 Antigen in 0.5 mL AS01B Adjuvant | Rabies Vaccine Rabipur
Started | 20 | 10
Completed | 19 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 50 ug of FMP010 Antigen in 0.5 mL AS01B Adjuvant: Plasmodium falciparum Malaria Protein 010 (FMP010): Vaccine antigen is a recombinant protein based on merozoite surface protein-1 (MSP-1) of FVO strain of Plasmodium falciparum, and adjuvant AS01B is a proprietary adjuvant of GSK
- Total: Total of all reporting groups
Arm/Group | 50 ug of FMP010 Antigen in 0.5 mL AS01B Adjuvant | Rabies Vaccine Rabipur | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 12 | 5 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 20 | 10 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Luo | 18 | 9 | 27
  Lulya | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Kenya | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events With Each Vaccination by Grade
Description: Vaccinations were given at 0-, 1-, 2-month interval, occurrence and intensity of solicited symptoms on day of vaccination (Day 0) and Days 1-7 after each vaccination Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe
Time Frame: After each vaccination (Day 0), follow-up visits were scheduled on Days 1, 2, 3, and 7
Measure: Count of Participants; unit: Participants
Groups:
- Rabies Vaccine Rabipur: Rabipur: Rabipur is a licensed rabies vaccine. Vaccinations were performed intramuscularly in the deltoid muscle of the non-dominant arm, 3 doses were given at 0-, 1-, 2-month interval.
Arm/Group | 50 ug of FMP010 Antigen in 0.5 mL AS01B Adjuvant | Rabies Vaccine Rabipur
Number analyzed (Participants) | 20 | 10
Participants
  Immunization 1: Fever: Grade 1 | 0 | 0
  Immunization 1: Fever: Grade 2 | 0 | 0
  Immunization 1: Fever: Grade 3 | 0 | 0
  Immunization 1: Fever: No experiences | 20 | 10
  Immunization 1: Fatigue: Grade 1 | 2 | 1
  Immunization 1: Fatigue: Grade 2 | 3 | 0
  Immunization 1: Fatigue: Grade 3 | 0 | 0
  Immunization 1: Fatigue: No experiences | 15 | 9
  Immunization 1: Gastrointestinal (nausea): Grade 1 | 3 | 1
  Immunization 1: Gastrointestinal (nausea): Grade 2 | 0 | 0
  Immunization 1: Gastrointestinal (nausea): Grade 3 | 0 | 0
  Immunization 1: Gastrointestinal (nausea): No experiences | 17 | 9
  Immunization 1: Headache: Grade 1 | 8 | 1
  Immunization 1: Headache: Grade 2 | 4 | 0
  Immunization 1: Headache: Grade 3 | 0 | 0
  Immunization 1: Headache: No experiences | 8 | 9
  Immunization 1: Malaise: Grade 1 | 2 | 0
  Immunization 1: Malaise: Grade 2 | 1 | 0
  Immunization 1: Malaise: Grade 3 | 0 | 0
  Immunization 1: Malaise: No experiences | 17 | 10
  Immunization 1: Myalgia: Grade 1 | 1 | 1
  Immunization 1: Myalgia: Grade 2 | 0 | 0
  Immunization 1: Myalgia: Grade 3 | 0 | 0
  Immunization 1: Myalgia: No experiences | 19 | 9
  Immunization 1: Joint pain: Grade 1 | 2 | 1
  Immunization 1: Joint pain: Grade 2 | 1 | 0
  Immunization 1: Joint pain: Grade 3 | 0 | 0
  Immunization 1: Joint pain: No experiences | 17 | 9
  Immunization 1: Local pain: Grade 1 | 14 | 6
  Immunization 1: Local pain: Grade 2 | 6 | 0
  Immunization 1: Local pain: Grade 3 | 0 | 0
  Immunization 1: Local pain: No experiences | 0 | 4
  Immunization: Local redness: Grade 1 | 1 | 0
  Immunization: Local redness: Grade 2 | 0 | 0
  Immunization: Local redness: Grade 3 | 0 | 0
  Immunization: Local redness: No experiences | 19 | 10
  Immunization 1: Local swelling: Grade 1 | 6 | 2
  Immunization 1: Local swelling: Grade 2 | 0 | 0
  Immunization 1: Local swelling: Grade 3 | 0 | 0
  Immunization 1: Local swelling: No experiences | 14 | 8
  Immunization 2: Fever: Grade 1 | 1 | 0
  Immunization 2: Fever: Grade 2 | 0 | 0
  Immunization 2: Fever: Grade 3 | 0 | 0
  Immunization 2: Fever: No experiences | 19 | 10
  Immunization 2: Fatigue: Grade 1 | 1 | 1
  Immunization 2: Fatigue: Grade 2 | 1 | 0
  Immunization 2: Fatigue: Grade 3 | 0 | 0
  Immunization 2: Fatigue: No experiences | 18 | 9
  Immunization 2: Gastrointestinal (nausea): Grade 1 | 0 | 0
  Immunization 2: Gastrointestinal (nausea): Grade 2 | 1 | 0
  Immunization 2: Gastrointestinal (nausea): Grade 3 | 0 | 0
  Immunization 2: Gastrointestinal (nausea): No experiences | 19 | 10
  Immunization 2: Headache: Grade 1 | 3 | 0
  Immunization 2: Headache: Grade 2 | 0 | 0
  Immunization 2: Headache: Grade 3 | 1 | 0
  Immunization 2: Headache: No experiences | 16 | 10
  Immunization 2: Malaise: Grade 1 | 2 | 0
  Immunization 2: Malaise: Grade 2 | 3 | 0
  Immunization 2: Malaise: Grade 3 | 0 | 0
  Immunization 2: Malaise: No experiences | 15 | 10
  Immunization 2: Myalgia: Grade 1 | 1 | 0
  Immunization 2: Myalgia: Grade 2 | 2 | 0
  Immunization 2: Myalgia: Grade 3 | 0 | 0
  Immunization 2: Myalgia: No experiences | 17 | 10
  Immunization 2: Joint pain: Grade 1 | 1 | 0
  Immunization 2: Joint pain: Grade 2 | 2 | 0
  Immunization 2: Joint pain: Grade 3 | 0 | 0
  Immunization 2: Joint pain: No experiences | 17 | 10
  Immunization 2: Local pain: Grade 1 | 12 | 5
  Immunization 2: Local pain: Grade 2 | 7 | 5
  Immunization 2: Local pain: Grade 3 | 0 | 0
  Immunization 2: Local pain: No experiences | 1 | 0
  Immunization 2: Local redness: Grade 1 | 3 | 2
  Immunization 2: Local redness: Grade 2 | 0 | 0
  Immunization 2: Local redness: Grade 3 | 0 | 0
  Immunization 2: Local redness: No experiences | 17 | 8
  Immunization 2: Local swelling: Grade 1 | 3 | 2
  Immunization 2: Local swelling: Grade 2 | 0 | 0
  Immunization 2: Local swelling: Grade 3 | 0 | 0
  Immunization 2: Local swelling: No experiences | 17 | 8
  Immunization 3: Fever: Grade 1 | 1 | 0
  Immunization 3: Fever: Grade 2 | 0 | 0
  Immunization 3: Fever: Grade 3 | 0 | 0
  Immunization 3: Fever: No experiences | 19 | 10
  Immunization 3: Fatigue: Grade 1 | 2 | 0
  Immunization 3: Fatigue: Grade 2 | 0 | 0
  Immunization 3: Fatigue: Grade 3 | 0 | 0
  Immunization 3: Fatigue: No experiences | 18 | 10
  Immunization 3: Gastrointestinal (nausea): Grade 1 | 0 | 0
  Immunization 3: Gastrointestinal (nausea): Grade 2 | 0 | 0
  Immunization 3: Gastrointestinal (nausea): Grade 3 | 0 | 0
  Immunization 3: Gastrointestinal (nausea): No experiences | 20 | 10
  Immunization 3: Headache: Grade 1 | 4 | 0
  Immunization 3: Headache: Grade 2 | 2 | 1
  Immunization 3: Headache: Grade 3 | 0 | 0
  Immunization 3: Headache: No experiences | 14 | 9
  Immunization 3: Malaise: Grade 1 | 1 | 0
  Immunization 3: Malaise: Grade 2 | 1 | 0
  Immunization 3: Malaise: Grade 3 | 0 | 0
  Immunization 3: Malaise: No experiences | 18 | 10
  Immunization 3: Myalgia: Grade 1 | 1 | 0
  Immunization 3: Myalgia: Grade 2 | 0 | 0
  Immunization 3: Myalgia: Grade 3 | 0 | 0
  Immunization 3: Myalgia: No experiences | 19 | 10
  Immunization 3: Joint pain: Grade 1 | 1 | 1
  Immunization 3: Joint pain: Grade 2 | 0 | 0
  Immunization 3: Joint pain: Grade 3 | 0 | 0
  Immunization 3: Joint pain: No experiences | 19 | 9
  Immunization 3: Local pain: Grade 1 | 10 | 4
  Immunization 3: Local pain: Grade 2 | 4 | 0
  Immunization 3: Local pain: Grade 3 | 0 | 0
  Immunization 3: Local pain: No experiences | 6 | 6
  Immunization 3: Local redness: Grade 1 | 0 | 0
  Immunization 3: Local redness: Grade 2 | 0 | 0
  Immunization 3: Local redness: Grade 3 | 1 | 0
  Immunization 3: Local redness: No experiences | 19 | 10
  Immunization 3: Local swelling: Grade 1 | 1 | 1
  Immunization 3: Local swelling: Grade 2 | 0 | 0
  Immunization 3: Local swelling: Grade 3 | 1 | 0
  Immunization 3: Local swelling: No experiences | 18 | 9

2. Primary Outcome: Number of Subjects With Unsolicited Adverse Events at Specified Grades
Description: Vaccinations were given at 0-, 1-, 2-month interval, number of subjects reporting unsolicited symptoms at specified grades over a 30-day follow-up period (day of vaccination and 29 subsequent days) after each vaccination
  Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe
Time Frame: After each vaccination (Day 0), 30 day f/u period post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 50 ug of FMP010 Antigen in 0.5 mL AS01B Adjuvant | Rabies Vaccine Rabipur
Number analyzed (Participants) | 20 | 10
Participants
  Grade 1 | 20 | 10
  Grade 2 | 15 | 9
  Grade 3 | 1 | 1

3. Primary Outcome: Number of Subjects With the Occurrence of Serious Adverse Events
Description: Vaccinations were given at 0-, 1-, 2-month interval, number of subjects with the occurrence of serious adverse events at days 0-7 post vaccination
Time Frame: After each vaccination (Day 0), follow-up visits were scheduled on Days 1, 2, 3, and 7 post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 50 ug of FMP010 Antigen in 0.5 mL AS01B Adjuvant | Rabies Vaccine Rabipur
Number analyzed (Participants) | 20 | 10
Participants | 0 | 0

4. Secondary Outcome: Antibody Titers Per Subject by Enzyme Linked Immunosorbent Assay in 50 µg Dose Group
Description: Antibody concentrations will be presented by reporting the summarized Geometric Mean Titer (GMT) values with 95% Confidence Interval (CI) (not presented in results), at each time point at which blood samples are taken for serology.
  Peak responses (Day 70) will be compared by Student's T test on data normalized by log transformation to ascertain presence or absence of significant dose response difference. GMTs are presented without CI data.
Time Frame: After each vaccination, blood draws performed on Days 0, 14, 28, 42, 56, 70 and 112
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | 50 ug of FMP010 Antigen in 0.5 mL AS01B Adjuvant
Number analyzed (Participants) | 20
Geometric Mean Titers
  Subject 00423: Day0 | 44720.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00423: Day14 | 54644.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00423: Day28 | 51390.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00423: Day42 | 97930.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00423: Day56 | 90560.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00423: Day70 | 99530.0 [NA to NA] — CICI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00423: Day112 | 91040.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00906: Day0 | 7055.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00906: Day14 | 7961.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00906: Day28 | 11322.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00906: Day42 | 36532.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00906: Day56 | 21780.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00906: Day70 | 36438.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 00906: Day112 | 14994.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02507: Day0 | 84830.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02507: Day14 | 261320.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02507: Day28 | 172340.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02507: Day42 | 224560.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02507: Day56 | 396580.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02507: Day70 | 275580.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02507: Day 112 | 240330.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02708: Day0 | 4905.9 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02708: Day14 | 7577.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02708: Day28 | 10519.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02708: Day42 | 61350.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02708: Day56 | 40838.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subect 02708: Day70 | 66650.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 02708: Day112 | 57170.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03401: Day0 | 2215.7 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03401: Day14 | 10186.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03401: Day28 | 6060.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03401: Day42 | 62353.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03401: Day56 | 30647.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03401: Day70 | 70680.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03401: Day112 | 45400.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03814: Day0 | 15190.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03814: Day14 | 45280.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03814: Day28 | 44100.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03814: Day42 | 83150.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03814: Day56 | 137740.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03814: Day70 | 80160.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 03814: Day112 | 99760.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 05029: Day0 | 4151.5 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 05029: Day14 | 15949.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 05029: Day28 | 21873.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 05029: Day42 | 92010.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 05029: Day56 | 58170.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 05029: Day70 | 74950.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 05029: Day112 | 41140.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06020: Day0 | 45960.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06020: Day14 | 45690.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06020: Day28 | 48483.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06020: Day42 | 65830.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06020: Day56 | 79880.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06020: Day70 | 68280.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06020: Day112 | 54958.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06627: Day0 | 3926.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06627: Day14 | 10662.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06627: Day28 | 8919.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06627: Day42 | 12677.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06627: Day56 | 10673.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06627: Day70 | 12201.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 06627: Day112 | NA [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 07722: Day0 | 399.6 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 07722: Day14 | 1500.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 07722: Day28 | 970.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 07722: Day42 | 55140.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 07722: Day56 | 39952.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 07722: Day70 | 127770.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 07722: Day112 | 40950.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08904: Day0 | 1751.8 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08904: Day14 | 2656.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08904: Day28 | 2176.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08904: Day42 | 19760.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08904: Day56 | 11798.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08904: Day70 | 16158.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08904: Day112 | 13393.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09105: Day0 | 37.7 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09105: Day14 | 567.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09105: Day28 | 1318.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09105: Day42 | 132810.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09105: Day56 | 37366.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09105: Day70 | 121030.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09105: Day112 | 30260.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09621: Day0 | 6147.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09621: Day14 | 15889.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09621: Day28 | 15213.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09621: Day42 | 32252.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09621: Day56 | 19676.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09621: Day70 | 53608.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09621: Day112 | 26482.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09913: Day0 | 29480.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09913: Day14 | 32260.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09913: Day28 | 27302.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09913: Day42 | 80040.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09913: Day56 | NA [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09913: Day72 | 76470.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09913: Day112 | 114600.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10015: Day0 | 2007.5 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10015: Day14 | 6241.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10015: Day28 | 6617.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10015: Day42 | 53650.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10015: Day56 | 311250.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10015: Day70 | 205460.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10015: Day112 | 149250.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10916: Day0 | 28200.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10916: Day14 | 53252.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10916: Day28 | 61407.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10916: Day42 | 68040.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10916: Day56 | 71610.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10916: Day70 | 60950.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10916: Day112 | 81650.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12217: Day0 | 6603.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12217: Day14 | 11804.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12217: Day28 | 10355.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12217: Day42 | 48342.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12217: Day56 | 24537.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12217: Day70 | 78190.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12217: Day112 | 45929.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12518: Day0 | 2051.6 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12518: Day14 | 4403.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12518: Day28 | 2214.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12518: Day42 | 78680.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12518: Day56 | 27675.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12518: Day70 | 126160.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12518: Day112 | 38900.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12612: Day0 | 1852.4 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12612: Day14 | 1545.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12612: Day28 | 979.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12612: Day42 | 7536.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12612: Day56 | 4067.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12612: Day70 | 23216.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12612: Day112 | 11960.0 [NA to NA] — CCI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 13209: Day0 | 940.8 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 13209: Day14 | 2506.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 13209: Day28 | 2988.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 13209: Day42 | 153550.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 13209: Day 56 | 900000.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 13209: Day70 | 110650.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 13209: Day112 | 38390.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure

5. Secondary Outcome: Antibody Titers Per Subject by Enzyme Linked Immunosorbent Assay in Rabies Vaccine Group
Description: Antibody concentrations will be presented by reporting the summarized Geometric Mean Titer (GMT) values with 95% Confidence Interval (CI) at each time point at which blood samples are taken for serology.
  Peak responses (Day 70) will be compared by Student's T test on data normalized by log transformation to ascertain presence or absence of significant dose response difference. GMTs are presented without CI data.
Time Frame: After each vaccination, blood draws performed on Days 0, 14, 28, 42, 56, 70 and 112
Measure: Mean (95% Confidence Interval); unit: Geometric Mean Titers
Arm/Group | Rabies Vaccine Rabipur
Number analyzed (Participants) | 10
Geometric Mean Titers
  Subject 01603: Day0 | 20580.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01603: Day14 | 23707.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01603: Day28 | 22537.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01603: Day42 | 24090.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01603: Day56 | 42005.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01603: Day70 | 43723.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01603: Day112 | 32104.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01702: Day0 | 71.5 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01702: Day14 | 84.3 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01702: Day28 | 53.2 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01702: Day42 | 57.8 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01702: Day56 | 65.1 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01702: Day70 | 73.6 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 01702: Day112 | 42.1 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04026: Day0 | 122.6 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04026: Day14 | 103.2 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04026: Day28 | 109.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04026: Day42 | 77.5 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04026: Day56 | 1000.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04026: Day70 | 544.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04026: Day112 | 125.8 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04328: Day0 | 5226.3 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04328: Day14 | 3782.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04328: Day28 | 4560.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04328: Day42 | 3788.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04328: Day56 | 2914.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04328: Day70 | 1920.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 04328: Day112 | 1802.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08725: Day0 | 27240.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08725: Day14 | 29477.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08725: Day28 | 26786.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08725: Day42 | 17866.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08725: Day56 | 13819.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08725: Day70 | 9601.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 08725: Day112 | 9898.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09211: Day0 | 2347.1 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09211: Day14 | 2250.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09211: Day28 | 2794.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09211: Day42 | 1952.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09211: Day56 | 1378.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09211: Day70 | 1232.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 09211: Day112 | 1991.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10324: Day0 | 3970.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10324: Day14 | 4493.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10324: Day28 | 3781.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10324: Day42 | 2891.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10324: Day56 | 3849.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10324: Day70 | 1901.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10324: Day112 | 1381.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10810: Day0 | 49410.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10810: Day14 | 41500.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10810: Day28 | 45920.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10810: Day42 | 49386.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10810: Day56 | 32158.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10810: Day70 | 39979.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 10810: Day112 | 36962.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 11819: Day0 | 9669.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 11819: Day14 | 11155.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 11819: Day28 | 10008.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 11819: Day42 | 9381.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 11819: Day56 | 6355.0 [NA to NA] — CCI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 11819: Day70 | 5276.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 11819: Day112 | 5921.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12330: Day0 | 1117.6 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12330: Day14 | 1291.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12330: Day28 | 1392.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12330: Day42 | 1105.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12330: Day56 | 734.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12330: Day70 | 858.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure
  Subject 12330: Day112 | 852.0 [NA to NA] — CI was not included in the tables section of the final clinical study report that corresponds to this outcome measure

ADVERSE EVENTS:
Time Frame: Day 0 - 146
Arm/Group | 50 µg of FMP010 Antigen in 0.5 mL AS01B Adjuvant | Rabies Vaccine Rabipur
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 19/20 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 µg of FMP010 Antigen in 0.5 mL AS01B Adjuvant (N=20) | Rabies Vaccine Rabipur (N=10)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abscesses on lower limbs (Infections and infestations) | 1 (1) | 0 (0)
Abscesses right medial malleolus (Infections and infestations) | 1 (1) | 0 (0)
Acute colitis (infective) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute gastroenteritis (amoebiasis) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Allergic conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Allergic conjunctivitis (both eyes) (Infections and infestations) | 1 (1) | 2 (2)
Allergic cough (Immune system disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Immune system disorders) | 1 (1) | 0 (0)
Allergic skin reaction (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis in both knee joints (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4)
Chest pain (musculoskeletal) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Chills and rigors (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (both eyes) (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (left eye) (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Decreased neutrophil count (Investigations) | 3 (3) | 0 (0)
Decreased white blood cell count (Investigations) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (6) | 2 (3)
Drop in hemoglobin (Investigations) | 1 (1) | 0 (0)
Drop in neutrophil count (Investigations) | 5 (5) | 5 (7)
Drop in platelet count (Investigations) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Elbow joint pain bilateral (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Elevated ALT (Investigations) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Entrocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye strain both eyes (Eye disorders) | 1 (1) | 0 (0)
Fullness of chest related heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fungal dermatitis (Infections and infestations) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
General body aches (General disorders) | 0 (0) | 1 (1)
General body weakness (General disorders) | 1 (1) | 0 (0)
Generalized joint pains (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized malaise (General disorders) | 1 (1) | 0 (0)
Giardiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 8 (14) | 3 (4)
Herpes labialis (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Hot flushes (Vascular disorders) | 1 (1) | 0 (0)
Hotness of body (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Itchiness of ears (mild) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itchiness of injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 2 (2) | 0 (0)
Loss of appetite (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Lumbago (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbosacral back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Malaria (Blood and lymphatic system disorders) | 9 (9) | 3 (3)
Mild cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mild drop in neutrophils (Investigations) | 1 (1) | 0 (0)
Muscular neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular pain lower back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neck pains (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Numbness left upper limb (Nervous system disorders) | 1 (1) | 1 (1)
Numbness of left arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Numbness of left arm (muscular) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pain at circumcision site (General disorders) | 1 (1) | 0 (0)
Pain both eyes (Eye disorders) | 1 (1) | 0 (0)
Pain left face (General disorders) | 1 (1) | 0 (0)
Pain on the left elbow joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain right shin (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (3) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus of the interphalangeal spaces, both feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus all over body (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Raised WBC count (Investigations) | 1 (1) | 0 (0)
Reduced appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Reduced neutrophil count (Investigations) | 0 (0) | 1 (1)
Relative eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Right chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right joint (hip) pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Small abscess left foot (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue injury left foot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue injury left heel (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury left shoulder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury right foot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue injury right hand (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury right wrist joint (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sore mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subjective fever (General disorders) | 2 (2) | 0 (0)
Subjective weakness of the left upper limb (Nervous system disorders) | 1 (1) | 0 (0)
Suidical ideations (Psychiatric disorders) | 0 (0) | 1 (1)
Tooth pain secodnary to dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth sensitivity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Torticollis (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 7 (10)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weakness of left arm (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No